CLINICAL TRIAL: NCT03651661
Title: Pupillographie Als Screeningtest für Cerebrale Insulinresistenz
Brief Title: Pupillography as Screening Tool for Brain Insulin Resistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 567/20168O2
Record Dates: First submitted 2018-07-02; First posted 2018-08-29 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2018-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Insulin

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nasal insulin (Active Comparator): 160 U of human insulin as nasal spray
  Interventions: Drug: human insulin; Diagnostic Test: Pupillography
- nasal placebo (Placebo Comparator): placebo as nasal spray
  Interventions: Drug: placebo; Diagnostic Test: Pupillography

INTERVENTIONS:
Drug: human insulin — human insulin administered as nasal spray
  Arms: nasal insulin
Drug: placebo — placebo administered as nasal spray
  Arms: nasal placebo
Diagnostic Test: Pupillography — Autonomic tone will be adressed by pupillography using the F2D2 (Amtech Germany) device.

SUMMARY:
Cerebral insulin action is important in the regulation of whole body glucose metabolism. However, the cerebral insulin action differs between individuals - there is a so called cerebral insulin resistance. The influence of central insulin action on peripheral metabolism seems at least partially mediated via the autonomous nervous system. A noninvasive method to measure autonomic function is the pupillography. The aim of the study is to find out whether pupillography can be used to assess central insulin activity. Thus, pupillography will be performed in 30 normal weight and 30 overweight subjects before and after application insulin intranasally.

ELIGIBILITY:
Inclusion Criteria:

* voluntary adults
* HbA1c <5.8%
* Age between 18 and 60 years
* written consent

Exclusion Criteria:

* There is a pregnancy or pregnancy can not be excluded
* lactating women
* Minors or non-consenting subjects are also excluded
* Acute illness or infection within the last 4 weeks
* Neurological and psychiatric disorders
* intake of centrally acting drugs
* Subjects with hemoglobin levels Hb <12g / dl (in females), Hb <14g / dl (males)
* Allergic diseases against one of the substances used

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2019-01-07 (Actual)

PRIMARY OUTCOMES:
Measurements of autonomic nervous system activity by pupillography | Measurements baseline and change to baseline 15 minutes and 30 minutes after spray application
  There will be measurements of autonomic nervous system activity by pupillography in order to identify central insulin action. The primary variable is the pupil width change in pupillography before compared to after intranasal insulin/placebo administration in 30 lean subjects. The investigation takes place in a darkened room with low backlight of about 5-10lx. The pupillographic recording is carried out with a commercially available device, F2D2 (Amtech Germany). In this case, the pupil width is recorded for 6 minutes continuously before and after nasal insulin (also 16 strokes of 10 E) or placebo doses with an infrared camera permanently mounted in a video goggle. Additionally, a possible change of the pupillary light reflection to monochromatic light is measured. Evaluation parameters are latency, amplitude and re-dilatation behavior.
Measurements of latency of pupil response to light stimulation. | Measurements baseline and change to baseline 15 minutes and 30 minutes after spray application
  There will be measurements of autonomic nervous system activity by pupillography in order to identify central insulin action. The investigation takes place in a darkened room with low backlight of about 5-10lx. The pupillographic recording is carried out with a commercially available device, F2D2 (Amtech Germany). A possible change of the pupillary light reflection to monochromatic light is measured. Evaluation parameter is latency. The responses before and after nasal spray administration will be compared.
Measurements of amplitude of pupil response to light stimulation. | Measurements baseline and change to baseline 15 minutes and 30 minutes after spray application
  There will be measurements of autonomic nervous system activity by pupillography in order to identify central insulin action. The investigation takes place in a darkened room with low backlight of about 5-10lx. The pupillographic recording is carried out with a commercially available device, F2D2 (Amtech Germany). A possible change of the pupillary light reflection to monochromatic light is measured. Evaluation parameter is amplitude . The responses before and after nasal spray administration will be compared.
Measurements of re-dilation behaviour of pupil response to light stimulation. | Measurements baseline and change to baseline 15 minutes and 30 minutes after spray application
  There will be measurements of autonomic nervous system activity by pupillography in order to identify central insulin action. The investigation takes place in a darkened room with low backlight of about 5-10lx. The pupillographic recording is carried out with a commercially available device, F2D2 (Amtech Germany). A possible change of the pupillary light reflection to monochromatic light is measured. Evaluation parameter is re-dilatation behavior. The responses before and after nasal spray administration will be compared.

SECONDARY OUTCOMES:
Autonomic nervous system | Measurements baseline and change to baseline 15 minutes and 30 minutes after spray application
  effect of nasal insulin or placebo spray on autonomic nervous system tone measured by heart rate variability.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tuebingen, Department of Internal Medicine IV, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No